CLINICAL TRIAL: NCT06412055
Title: Optimizing Gait with Bidirectional Tuning of the Ankle-foot Orthosis (AFO) Stiffness in People with Lower Leg Muscle Weakness
Brief Title: Bidirectional Tuning of the AFO Stiffness
Acronym: NEUROSWING
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: FIOR & GENTZ (Unknown)
Responsible Party: Principal Investigator, Merel Brehm, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL85684.018.23
Record Dates: First submitted 2024-05-02; First posted 2024-05-14 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Neuromuscular Disorders
Keywords: Neuromuscular disorders; dorsiflexor and plantarflexor weakness; ankle-foot orthosis (AFO); bidirectional stiffness tuning; Gait kinetics and kinematics; Walking energy cost; Perceived physical functioning
MeSH Terms: conditions — Neuromuscular Diseases

STUDY DESIGN:
Intervention Model Description: pilot self-controlled intervention study with measurements of three spring-like AFOs (WalkOn Reaction® (Ottobock, Duderstadt), the Matrix Max2® (TruLife, Dublin, Ireland), and the Matrix® (TruLife, Dublin, Ireland)) having the same stiffness in both directions, and a newly custom-made spring-hinged AFO with the NEURO SWING® system ankle joint with individualized spring settings (Fior& Gentz, Lüneburg, Germany) directly after delivery and 6 weeks post-delivery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- NEURO SWING AFO (Experimental): Participants will be fitted with a new custom-made spring-hinged AFO with the NEURO SWING® system ankle joint. Following a previously developed algorithm, the stiffness will be individually selected from six different configurations tested during an optimization measurement directly after delivery of the new AFO. Thereafter, participants will use the optimized AFO with individualized stiffness at home for six weeks during the course of the study.
  Interventions: Device: NEURO SWING AFO (Fior& Gentz, Lüneburg, Germany); Device: WalkOn Reaction® (Ottobock, Duderstadt); Device: Matrix Max2® (TruLife, Dublin, Ireland); Device: Matrix® (TruLife, Dublin, Ireland)

INTERVENTIONS:
Device: NEURO SWING AFO (Fior& Gentz, Lüneburg, Germany) — stiffness-optimized custom-made spring-hinged AFO with the NEURO SWING® system ankle joint build in
Device: WalkOn Reaction® (Ottobock, Duderstadt) — comparator: prefab spring-like AFO without hinge with a predefined stiffness (2.8 Nm/degree).
Device: Matrix Max2® (TruLife, Dublin, Ireland) — comparator: prefab spring-like AFO without hinge with a predefined stiffness (1.4 Nm/degree)
Device: Matrix® (TruLife, Dublin, Ireland) — comparator: prefab spring-like AFO without hinge with a predefined stiffness (0.6 Nm/degree)

SUMMARY:
The goal of this pilot study with a pre-post design is to investigate the effects of separate individualization of the AFO stiffness towards plantar- and dorsiflexion in a spring-hinged AFO on walking compared to a spring-like AFO (3 types) having the same stiffness in both directions.

People with a neuromuscular disease or nerve injury causing at least plantarflexor weakness (determined as the inability to perform 3 single heel rises), with an indication for or using an AFO, will be fitted with a new, custom-made spring-hinged AFO with the NEURO SWING® system ankle joint (Fior& Gentz, Lüneburg, Germany), of which the stiffness of ventral and dorsal compartment of this spring-hinged AFO will be individualized. For comparison, measurements will be performed with three different prefab spring-like AFOs with different stiffness levels (but which have a similar stiffness towards plantar and dorsiflexion), and the participants' current AFO if applicable, and shoes-only at baseline.

The main outcome parameters will be the maximal ankle plantarflexion angle, ankle angular velocity and knee flexion angle during the loading response, which will be measured using a 3D gait analysis. Secondary outcomes include other gait biomechanics, walking energy cost, walking speed, standing balance, perceived physical functioning and perceived walking ability.

DETAILED DESCRIPTION:
Many neuromuscular diseases cause weakness of the ankle dorsiflexors and plantarflexors, resulting in an altered gait pattern. In particular, weakness of the plantar flexors leads to a reduced walking ability as it hampers safety in both standing and walking. The primary treatment to improve walking ability and safety during standing and walking in dorsiflexor and/or plantarflexor weakness is the provision of ankle-foot orthoses (AFOs). To maximize treatment outcomes in case of lower leg weakness, the optimal AFO stiffness needs to be individually determined. Individual optimization of the stiffness can be performed with a spring-like AFO or with a spring-hinged AFO. With a spring-like AFO, the stiffness towards plantar- and dorsiflexion is similar, oftentimes resulting in a higher than necessary stiffness towards plantarflexion. An advantage of spring-hinged AFOs is that, unlike spring-like AFOs, the stiffness can be separately optimized in the directions of dorsiflexion and plantarflexion.

The objective of this pilot study is to evaluate the effects of separate individualization of the AFO stiffness towards plantar- and dorsiflexion in a spring-hinged AFO compared to three types of spring-like AFO having the same stiffness in both directions on gait biomechanics, walking energy cost, walking speed, and standing balance. Additionally, effects will be evaluated of the optimal spring-hinged AFO 6 weeks after delivery of the AFO on perceived physical functioning, walking ability and satisfaction in daily life compared to the participants' AFO used at baseline if applicable or walking with shoes-only.

In this pilot study with a pre-post design, people with a neuromuscular disease or nerve injury causing at least plantarflexor weakness with an indication for or using an AFO will be fitted with a new, custom-made spring-hinged AFO with the NEURO SWING® system ankle joint (Fior& Gentz, Lüneburg, Germany). The stiffness of ventral and dorsal compartment of this spring-hinged AFO will be individualized using a previously developed optimization algorithm. The spring-hinged AFO with optimal stiffness settings will be used at home for 6-weeks. For comparison, the investigators will test the direct effects of three different prefab spring-like AFOs with different stiffness levels (but which have a similar stiffness towards plantar and dorsiflexion) of 2.8, 1.4 and 0.6 Nm/degrees respectively in a randomized order, and the participants' current AFO if applicable, and shoes-only at baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older;
2. Presence of plantar flexor weakness in at least one leg, determined as a score lower than 5 on the manual muscle testing scale (Medical Research Council- MRC) and/or inability to perform three single heel rises, with or without dorsiflexion weakness;
3. Indicated for or using an AFO;
4. Ability to walk 6-minutes consecutively (with assistive device, if necessary).

Exclusion Criteria:

1. When wearing the AFO, not able to walk short bouts of 10m without walking aids, such as a walker;
2. Foot deformities that do not fit in prefab spring-like AFOs;
3. Weakness of the knee extensor muscles, for which a knee-ankle-foot orthosis is indicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
maximal ankle angular velocity in loading response in degrees | day 0 (directly post-delivery)
  measured during a 3D gait analysis

SECONDARY OUTCOMES:
maximal ankle angular velocity in loading response | 6 weeks post-delivery for the stiffness-optimized NEURO SWING AFO
  measured during a 3D gait analysis
minimal ankle angle in loading response in degrees | day 0 (directly post-delivery) and 6 weeks post-delivery for the stiffness-optimized NEURO SWING AFO only
  measured during a 3D gait analysis
ankle angle during midstance in degrees | day 0 (directly post-delivery) and 6 weeks post-delivery for the stiffness-optimized NEURO SWING AFO only
  measured during a 3D gait analysis
maximal ankle angle during the stance phase in degrees | day 0 (directly post-delivery) and 6 weeks post-delivery for the stiffness-optimized NEURO SWING AFO only
  measured during a 3D gait analysis
maximal ankle moment in Nm/kg | day 0 (directly post-delivery) and 6 weeks post-delivery for the stiffness-optimized NEURO SWING AFO only
  measured during a 3D gait analysis
maximal ankle push-off power in Watt/kg | day 0 (directly post-delivery) and 6 weeks post-delivery for the stiffness-optimized NEURO SWING AFO only
  measured during a 3D gait analysis
maximal knee flexion angle in loading response in degrees | day 0 (directly post-delivery) and 6 weeks post-delivery for the stiffness-optimized NEURO SWING AFO only
  measured during a 3D gait analysis
minimal knee flexion angle during the stance phase in degrees | day 0 (directly post-delivery) and 6 weeks post-delivery for the stiffness-optimized NEURO SWING AFO only
  measured during a 3D gait analysis
maximal external knee flexion moment in loading response in degrees | day 0 (directly post-delivery) and 6 weeks post-delivery for the stiffness-optimized NEURO SWING AFO only
  measured during a 3D gait analysis
minimal external knee flexion moment during the stance phase in Nm/kg | day 0 (directly post-delivery) and 6 weeks post-delivery for the stiffness-optimized NEURO SWING AFO only
  measured during a 3D gait analysis
maximal hip power during loading response in Watt/kg | day 0 (directly post-delivery) and 6 weeks post-delivery for the stiffness-optimized NEURO SWING AFO only
  measured during a 3D gait analysis
maximal hip power during ankle push-off in Watt/kg | day 0 (directly post-delivery) and 6 weeks post-delivery for the stiffness-optimized NEURO SWING AFO only
  measured during a 3D gait analysis
walking speed in m/s | day 0 (directly post-delivery) and 6 weeks post-delivery for the stiffness-optimized NEURO SWING AFO only
  Walking speed will be measured during a 6-minute walk test (6MWT) at a self-selected comfortable speed.
walking energy cost in J/kg/m | day 0 (directly post-delivery) and 6 weeks post-delivery for the stiffness-optimized NEURO SWING AFO only
  During a 6-minute walk test (6MWT) at comfortable speed, oxygen uptake (VO2) and carbon dioxide production (VCO2) will be measured using a breath-by-breath gas analysis system (K5, Cosmed, Rome, Italy) worn on the patient's back. Over at least one minute during the last three minutes of the test, walking energy cost will be calculated from these measured parameters and the comfortable walking speed.
velocity of center-of-pressure displacement in mm/s | day 0 (directly post-delivery) and 6 weeks post-delivery for the stiffness-optimized NEURO SWING AFO only
  During the 3D gait analysis, a standing balance test will be performed. Participants will stand on one force plate with a standardised distance of 10 cm between the medial borders of the feet for 30 seconds. Standing posture, in terms of joint angles, will be determined using the markers placed according to the Plug-in-Gait model. Postural sway will be calculated as the Center-of-Pressure displacement during the last 15 seconds of the test.
center-of-pressure displacement in mm | day 0 (directly post-delivery) and 6 weeks post-delivery for the stiffness-optimized NEURO SWING AFO only
  During the 3D gait analysis, a standing balance test will be performed. Participants will stand on one force plate with a standardised distance of 10 cm between the medial borders of the feet for 30 seconds. Standing posture, in terms of joint angles, will be determined using the markers placed according to the Plug-in-Gait model. Postural sway will be calculated as the Center-of-Pressure displacement during the last 15 seconds of the test.
Perceived walking ability | baseline and 6 weeks post-delivery of the stiffness-optimized NEURO SWING AFO
  Perceived walking ability in terms of satisfaction, intensity, safety and stability during walking will be measured on a 10-point Numerical Rating Scale (NRS) ranging from 0 (worst possible score) to 10 (best possible score).
Perceived physical functioning | baseline and 6 weeks post-delivery of the stiffness-optimized NEURO SWING AFO
  Physical functioning will be measured using the physical functioning scale of the 36-item short form health survey (SF-36), with range 0-100 (a higher score means a better functioning).

OTHER OUTCOMES:
number of participants with adverse events | from baseline to 6 weeks post-delivery of the stiffness-optimized NEURO SWING AFO
  Adverse events are defined as any undesirable experience occurring to a subject during the study, whether or not considered related to the investigational product or experiments. The following adverse events reported spontaneously by the subject or observed by the investigator or his staff will be recorded; pressure sores, muscle soreness, pain, and falls.

CONTACTS AND LOCATIONS:
Overall Officials: Frans Nollet, MD PhD, Study Director — Amsterdam UMC, location AMC
Locations (1):
- Department of rehabilitation medicine Amsterdam UMC, location AMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data (IPD) and meta data will be made available to third parties via Figshare. Other anonymized IPD and documents will be made available on request including data analyses codes such as SPSS syntaxes.